CLINICAL TRIAL: NCT05488743
Title: Youth Smoking Prevention Program in Poland
Brief Title: Smoking Prevention Program in Poland
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Wroclaw Medical University (Other)
Collaborators: Stanford Reach Lab - Tobacco Prevention Toolkit (Unknown); American Association for Cancer Education (Unknown)
Responsible Party: Principal Investigator, Łukasz Moskal, MD, Principal Investigator, Wroclaw Medical University
Other Study IDs: Smoking Prevention
Record Dates: First submitted 2022-07-29; First posted 2022-08-05 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Smoking; Smoking Behaviors; Smoking (Tobacco) Addiction; E-cigarette Use; Vaping
Keywords: tobacco prevention cancer; smoking prevention; cancer education; educational intervention; cardiovascular diseases prevention; youth
MeSH Terms: conditions — Smoking; Behavior, Addictive; Vaping | interventions — Early Intervention, Educational

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 7th and 8th grade students (children age 12-15 years) from the elementary school
  Interventions: Behavioral: educational intervention

INTERVENTIONS:
Behavioral: educational intervention — The program consists of five 50-minutes sessions conducted in person as scheduled during weekly class meetings. Educators will conduct workshops with PowerPoint presentations and worksheets dedicated to in-class activities.

SUMMARY:
Smoking Prevention Program is a pilot exploratory study with a standardized curriculum based on the Tobacco Prevention Toolkit from Stanford University and translated into Polish by the members of Students Scientific Association of Oncology at Wroclaw Medical University. The program will assess the effectiveness of a school-based smoking prevention curricula keeping children as never smokers and test the feasibility of engaging medical students and teachers in implementing and evaluating a validated program on smoking prevention within the Polish School System. The research protocols, methods and data collection instruments of a standardized classroom based valid tobacco prevention program from Stanford University will be used for the study. The smoking prevention program is centred on drug resistance, personal self-management and increasing social skills. The program increases knowledge and uses coaching and practice to provide students with the skills to resist social pressures around cigarette use. The secondary outcome of this study is to determine the change in attitudes by Polish Medical Student regarding Cancer Prevention Research. During Smoking Prevention Program workshops, the 5-Session Curriculum for primary schools will be translated, applied and evaluated for polish students.

This community-based pilot will engage medical students, the local school district and the local health authority. The Educational program meets the requirements set by Centers for Disease Control and Prevention (CDC) in Guidelines for School Health Programs to Prevent Tobacco Use and Addiction. Following parental consent, the program will be implemented with all 7th and 8th grade students (children age 12-15 years) from the Elementary School in Tyniec Mały. This project is supported by the Head of Lower Silesian Oncology Center, the Head of Department of Oncology of Wroclaw Medical University, the Health and Social Affairs Department of City of Wroclaw and under the patronage of the Lower Silesia Governor's Office, the Polish Society of Oncology, the Polish Society of Public Health, the Lower Silesian Department of Polish Society of Cardiology and the European Association for Cancer Education (EACE).

Smoking Prevention Program is funded by the READS Grant Program from the American Association for Cancer Education (AACE).

ELIGIBILITY:
Inclusion Criteria:

* Students from Tyniec Mały
* 7th and 8th graders of the elementary school
* Parental consent
* Students consent

Exclusion Criteria:

* Lack of parental consent
* Lack of students consent

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The program will be implemented with all 7th and 8th grade students (children age 12-15 years) from the Elementary School in Tyniec Mały.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-08-13 (Estimated); Study Completion 2022-10-14 (Estimated)

PRIMARY OUTCOMES:
Smoking intention | 2 months
  Change in smoking intention among elementary school students after program completion (score based on survey results).
Knowledge of negative consequences of smoking | 2 months
  Change in knowledge about adverse effects of smoking after program completion (score based on survey results).

CONTACTS AND LOCATIONS:
Overall Officials: Łukasz Moskal, MD, Principal Investigator — Wroclaw Medical University; Konrad Reszka, MD, Principal Investigator — Wroclaw Medical University; Urszula Staszek-Szewczyk, MD, PhD, Principal Investigator — Wroclaw Regional Comprehensive Cancer Center, Department of Brachytherapy; Jagoda Łaba, MD, Principal Investigator — Wroclaw Medical University; Krzysztof Szewczyk, MD, PhD, Principal Investigator — Wroclaw Medical University, Department of Oncology, Division of Surgical Oncology
Locations (1):
- Wroclaw Medical University, Wroclaw, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Birge M, Duffy S, Miler JA, Hajek P. What Proportion of People Who Try One Cigarette Become Daily Smokers? A Meta-Analysis of Representative Surveys. Nicotine Tob Res. 2018 Nov 15;20(12):1427-1433. doi: 10.1093/ntr/ntx243. PMID 29126298
- [Background] Kaleta D, Polanska K, Rzeznicki A, Stelmach W, Wojtysiak P. Tobacco use patterns, knowledge, attitudes towards tobacco and availability of tobacco control training among school personnel from a rural area in Poland. Tob Induc Dis. 2017 Jan 11;15:3. doi: 10.1186/s12971-016-0110-y. eCollection 2017. PMID 28096794
- See also: World Health Organization. Regional Office for Europe. 2020. Summary results of the global youth tobacco survey in selected countries of the WHO European Region. World Health Organization. Regional Office for Europe. — http://apps.who.int/iris/bitstream/handle/10665/336752/WHO-EURO-2020-1513-41263-56157-eng.pdf?sequence=1&isAllowed=y